CLINICAL TRIAL: NCT06835647
Title: Maternal Fetal Device Performance Testing During Antepartum Twin Monitoring
Brief Title: Maternal Fetal Device Performance Twins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SA-000073
Record Dates: First submitted 2025-02-11; First posted 2025-02-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy
Keywords: Pregnancy; Twins

STUDY DESIGN:
Intervention Model Description: Pregnant women of ≥30 0/7 weeks gestation will undergo one 40-minute monitoring session utilizing the investigational device with two Doppler transducers (FHR 1 and FHR 2) following M- mode fetal ultrasound imaging confirming fetal presentation (i.e. vertex, breech, shoulder), fetal lie (i.e. longitudinal, transverse), visualization of fetal heart rates of each fetus and documentation. During the monitoring sessions, maternal pulse rate (MPR) will be monitored using a SpO2 sensor and the investigator shall be present to adjust the transducers as needed to maintain a continuous FHR tracing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Twin Monitoring - All Subjects (Experimental): Pregnant women of ≥30 0/7 weeks gestation will undergo one 40-minute monitoring session utilizing the investigational device with two Doppler transducers (FHR 1 and FHR 2) following M- mode fetal ultrasound imaging confirming fetal presentation, fetal lie, visualization of fetal heart rates of each fetus and documentation. During the monitoring sessions, maternal pulse rate (MPR) will be monitored using a SpO2 sensor and the investigator shall be present to adjust the transducers as needed to maintain a continuous FHR tracing.
  Interventions: Device: Investigational Fetal Monitor; Device: Ultrasound Imaging Device

INTERVENTIONS:
Device: Investigational Fetal Monitor — Investigational Fetal Monitoring Device Device is a multi-parameter maternal fetal monitor that is intended to monitor, store, display, transmit, and generate alarms for non-invasive and invasive clinical parameters of pregnant women and fetuses (singleton and twin), during the antepartum, intrapartum, and postpartum period.
Device: Ultrasound Imaging Device — The Ultrasound imaging device is a general-purpose diagnostic ultrasound system for use in measurement, display and analysis of the human body and fluid.

SUMMARY:
Maternal Fetal Monitoring devices assist the health care professional in acquiring, monitoring, and storing fetal and maternal physiologic data which support clinical decision making for pregnant women and assesses the overall fetal health status during pregnancy and delivery. This study aims to support a new maternal fetal monitoring device with clinical data by collecting simultaneous, continuous, external, distinguishable FHRs from twin pregnancies using ultrasound Doppler transducers from the new maternal fetal monitoring investigational device and a marketed ultrasound imaging device.

DETAILED DESCRIPTION:
This study aims to support a new maternal fetal monitoring device with clinical data by collecting distinguishable FHRs from twin pregnancies using ultrasound Doppler transducers from the investigational device and a marketed ultrasound imaging device. This study will collect twin fetal heart rate data from the new monitor on twin gestations.

Funding for this study will be provided by GE HealthCare. This study does not include patient advisors.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Twin pregnancy.
3. Aged 18+.
4. Greater than or equal to 30 0/7 weeks gestation.
5. Patient has none of the exclusion criteria.

Exclusion Criteria:

1. Non-twin pregnancy.
2. Involvement in another clinical trial currently or previously in this pregnancy that, in the investigator's opinion, would affect the conduct of this study.
3. Medical or obstetric problem that in investigator's opinion would make the patient incapable of taking part in the study.
4. Inability to understand the consent information due to medical illness, diminished intellectual capacity, or insurmountable language barrier.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of Distinct Fetal Heart Rate | 40 minutes
  Collection of simultaneous, distinct fetal heart rate from SpO2 data from one investigational device over a 40 minutes of continuous fetal monitoring.
Collection of Maternal Pulse Rate | 40 minutes
  Collection of maternal pulse rate from SpO2 data from one investigational device over a 40 minutes of continuous fetal monitoring.

SECONDARY OUTCOMES:
Incidence of Safety Events | 4 months
  Analysis of adverse events will be listed per subject, summarized with counts and percentages of events, and summarized with counts and percentages of subjects with events.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, NP, Principal Investigator — Element Materials Technology
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulrich CC, Dewald O. Pregnancy Ultrasound Evaluation(Archived). 2023 Feb 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557572/ PMID 32491504
- [Background] Euliano TY, Darmanjian S, Nguyen MT, Busowski JD, Euliano N, Gregg AR. Monitoring Fetal Heart Rate during Labor: A Comparison of Three Methods. J Pregnancy. 2017;2017:8529816. doi: 10.1155/2017/8529816. Epub 2017 Mar 14. PMID 28392944
- [Background] Andelija S, Tafti D. Sonography Fetal Assessment, Protocols, and Interpretation. 2023 May 22. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK576427/ PMID 35015452